CLINICAL TRIAL: NCT03855917
Title: A Phase IV Open-label Multicentre International Pilot Study of 4-week Treatment With Sofosbuvir (400 mg) Plus Glecaprevir/Pibrentasvir (300mg/120mg) in Chronic HCV Treatment naïve Patients With Early Liver Disease
Brief Title: Strategic Treatment Reduction in Very Early Liver Disease With 4 Weeks Sofosbuvir Plus Glecepravir-pibrentasvir
Acronym: STRIVE-4
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHCRP1901
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; glecaprevir; pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sof plus G/P (Experimental): Four weeks of sofosbuvir (400mg) plus glecaprevir-pibrentasvir (300mg/120mg) will be administered, followed by immediate retreatment of virological relapse with glecepravir/pibrentasvir (300mg/120mg) for 12 weeks, in treatment-naïve participants with chronic HCV infection and early liver disease (F0-F2).
  Interventions: Drug: Sofosbuvir 400mg [Sovaldi]; Drug: Glecaprevir/pibrentasvir (300mg/120mg)

INTERVENTIONS:
Drug: Sofosbuvir 400mg [Sovaldi] — Four weeks.
  Other Names: Sovaldi
Drug: Glecaprevir/pibrentasvir (300mg/120mg) — Four weeks.
  Other Names: Maviret

SUMMARY:
This study aims to evaluate the efficacy, safety and feasibility of four weeks of sofosbuvir plus glecaprevir-pibrentasvir, followed by immediate retreatment of virological relapse with glecepravir-pibrentasvir for 12 weeks, in treatment-naïve participants with chronic HCV infection and early liver disease (F0-F2).

DETAILED DESCRIPTION:
The capacity to eliminate HCV through rapid direct acting antiviral (DAA) therapy scale-up would be enhanced by shortened duration therapy in key populations. The "next generation" DAA regimen of glecaprevir/pibrentasvir (300mg/120mg), an NS3/4a protease inhibitor and NS5A inhibitor, provides key features for potential simplified shortened duration therapy in people with early liver disease (F0-2), including pangenotypic activity, high efficacy, and favourable on-treatment HCV RNA kinetics. The addition of sofosbuvir (400 mg) may provide further feasibility for shortened duration therapy with a potent triple class DAA regimen.

Shortened duration therapy (4-6 weeks) has been evaluated in chronic HCV populations with several DAA regimens, with generally unfavourable outcomes (SVR<50%) for 4 week durations.8-11 In a study among a predominantly African American population of 4 week duration therapy of 3 or 4 DAAs, with sofosbuvir/ledipasvir/GS-9451 (protease inhibitor) and sofosbuvir/ledipasvir/GS-9451/GS-9669 (non-nucleoside polymerase inhibitor), SVR was only 40% (10/25) and 20% (5/25) in the 3 and 4 DAA regimen groups, respectively.10 In separate phase II studies that included evaluation of 6 weeks sofosbuvir (400mg)/velpatasvir (100mg)/voxilaprevir (100 mg) in treatment naïve patients without cirrhosis, SVR was 88% (29/33) among patients with genotype 2, 3, 4, or 6,12 93% (14/15) in patients with genotype 13,13 and and 71% (24/34) in patients with genotype 1.14 Non-published data (provided by Gilead Sciences) from the latter study demonstrates a higher SVR (88%, 14/16) in the sub-population of patients with F0-2. Thus, in patients with relatively early liver disease virological failure is uncommon with 6-week duration sofosbuvir/velpatasvir/voxilaprevir therapy.

These studies would suggest that a 6-week duration therapy, particularly with a potent 3 DAA triple class regimen, may be feasible for many patients with chronic HCV infection, but a 4-week duration would probably compromise treatment outcomes. However, in a small study (n=16) among younger people who inject drugs (PWID) with early liver disease (<50 years, F0-2) in Denmark, a 4-week regimen of sofosbuvir/ledipasvir plus ribavirin provided a per protocol (PP)(n=13) SVR of 92% (one relapse) with intention to treat (ITT) SVR of 75%. In the same study 16 PWID were treated with the same regimen plus pegylated interferon with PP and ITT SVR of 100% and 94%, respectively. Further evidence for the potential of ultra-short duration DAA therapy comes from a response-guided study in Hong Kong. Patients with HCV genotype 1b were treated with three different triple class DAA regimens, including sofosbuvir/ledipasvir + asunaprevir, sofosbuvir + daclatasvir + simeprevir, or sofosbuvir + daclatasvir + asunaprevir, and those with an ultra-rapid virological response (HCV RNA <500 IU/mL at day 2; 18/26) had treatment duration shortened to three weeks. The SVR rate was 100% (18/18) in the three-week treated population.

While efficacy has been suboptimal in most studies of short duration DAA therapy to date, the emergence of clinically significant resistance-associated substitutions (RAS) has not been seen, and retreatment with the same regimen for 12 weeks has been successful.8,9 The FOURward study examined the safety and efficacy of short-duration therapy (4 or 6 weeks) with sofosbuvir + daclatasvir/asunaprevir/beclabuvir in patients with HCV genotype 1 and without cirrhosis.9 Although efficacy was suboptimal (SVR12 43%), among those with virological relapse (n=16), 44% (n=7) had no emergent RAS detected at failure. Furthermore, in the nine patients with treatment-emergent NS5A RAS, the clinical significance was uncertain, as all emergent NS5A RAS conferred low-nanomolar resistance in vitro. Regardless of RAS emergence, retreatment of patients who experienced virological relapse with 12 weeks sofosbuvir + daclatasvir/asunaprevir/beclabuvir + ribavirin resulted in SVR of 100%. C-SWIFT evaluated the efficacy and safety of sofosbuvir + elbasvir/grazoprevir in patients with HCV genotype 1 and without cirrhosis for four and six weeks, with SVR12 rates of 32% (10/31) and 87% (26/30), respectively.8 All patients with virological relapse who received retreatment with 12 weeks of sofosbuvir + elbasvir/grazoprevir + ribavirin achieved SVR12, despite the majority having NS5A and/or NS3 RAS.

The combination of sofosbuvir (400 mg) + glecaprevir/pibrentasvir (300mg/120mg) has not been evaluated as a shortened duration triple class DAA regimen. It has been evaluated as a 12 and 16-week regimen in combination with ribavirin for treatment of prior glecaprevir-pibrentasvir virological failure (8 or 12-week duration prior therapy), with very high efficacy of 96% (22/23) and good tolerability (Wyles D. et al. ILC 2018). A non-ribavirin containing regimen would be expected to have further enhanced tolerability.

ELIGIBILITY:
Inclusion Criteria:

- Participants must meet all inclusion criteria to be eligible to participate in this study:

1. Have voluntarily signed the informed consent form.
2. 18 years of age or older.
3. Chronic HCV infection as defined by anti-HCV antibody or HCV RNA detection for greater than 6 months.
4. Quantifiable HCV RNA at screening.
5. HCV treatment naïve (no prior treatment with an approved or investigation anti-HCV medication).
6. Liver fibrosis stage F0-F2, defined by at least one of the following:

   1. Liver stiffness measurement <9.5 kPa by transient elastography (FibroScan®)
   2. AST to platelet ratio index (APRI) <0.5
   3. Liver biopsy
7. If co-infection with HIV is documented, the subject must meet the following criteria:

   * ART naïve with CD4 T cell count >500 cells/mm3; OR
   * On a stable ART regimen (containing only permissible ART - see protocol section 6.3) for >8 weeks prior to screening visit, with CD4 T cell count >200 cells/mm3 and a plasma HIV RNA level below the limit of detection.
8. Negative pregnancy test at screening and baseline (females of childbearing potential only).
9. All fertile females must be using effective contraception during treatment and during the 30 days after treatment end.

Exclusion Criteria:

* Participants who meet any of the exclusion criteria are not to be enrolled in this study.

  1. History of any of the following:

     1. Clinically significant illness (other than HCV) or any other major medical disorder that may interfere with the participant treatment, assessment or compliance with the protocol; participants currently under evaluation for a potentially clinically significant illness (other than HCV) are also excluded.
     2. Clinical hepatic decompensation (i.e. ascites, encephalopathy or variceal haemorrhage).
     3. Solid organ transplant.
     4. History of severe, life-threatening or other significant sensitivity to any excipients of the study drugs.
  2. Any of the following lab parameters at screening:

     1. ALT > 10 x ULN
     2. AST > 10 x ULN
     3. Direct bilirubin > ULN
     4. Platelets < 150,000/μL (cells/mm3)
     5. Creatinine clearance (CLcr) < 50 mL/min
     6. Albumin < LLN
     7. INR > 1.5 ULN
  3. Pregnant or breastfeeding female.
  4. HBV infection (HBsAg positive).
  5. Use of prohibited concomitant medications as described in protocol section 6.3.
  6. Chronic use of systemically administered immunosuppressive agents (e.g. prednisone equivalent > 10 mg/day for >2 weeks).
  7. Therapy with any anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) ≤6 months prior to the first dose of study drug.
  8. Any investigational drug ≤6 weeks prior to the first dose of study drug.
  9. Ongoing severe psychiatric disease as judged by the treating physician.
  10. Inability or unwillingness to provide informed consent or abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
SVR12 | 16 weeks
  To evaluate the proportion achieving a sustained virological response at 12 weeks post treatment (SVR12) with sofosbuvir (400 mg) plus glecaprevir/pibrentasvir (300mg/120mg) for four weeks.

SECONDARY OUTCOMES:
Virological relapse | 16 weeks
  To evaluate virological relapse following 4 weeks sofosbuvir (400 mg) plus glecaprevir/pibrentasvir (300mg/120mg) in HCV treatment-naïve chronic HCV patients with early liver disease (F0-2).
Relapse characteristics | 32 weeks
  In patients with virological relapse, to evaluate the time course of relapse and emergence of treatment-associated resistance substitutions.
Re-treatment SVR | 32 weeks
  To evaluate SVR following re-treatment of virological relapse with 12 weeks glecaprevir/pibrentasvir (300mg/120mg).
Adherence | 32 weeks
  To evaluate the proportion adherent to treatment and study visits.
Cost-effectiveness | 32 weeks
  To evaluate cost-effectiveness of a shortened duration with re-treatment of relapse strategy, against a standard duration (8-week, historical data).

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Martinello, MD, PhD, Principal Investigator — Kirby Institute
Locations (3):
- Australia (3):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Blacktown Mt Druitt Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No
Protocol and SAP will be submitted along with the primary manuscript for publication.